CLINICAL TRIAL: NCT00656422
Title: Weight Gain, Eating Patterns, and Development of Body Composition During Initiation of Basal Insulin Therapy in Patients With Type 2 Diabetes: A Comparison of Insulin Detemir and Insulin Glargine
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Collaborators: Medical University of Vienna (Other); University of Bern (Other); CenTrial GmbH (Industry)
Responsible Party: University Hospital of Tübingen, Medical Department
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: N-ISP-1; LEV-002
Record Dates: First submitted 2008-04-04; First posted 2008-04-11 (Estimated); Last update posted 2012-11-01 (Estimated); Status verified 2012-10

CONDITIONS: Diabetes; Obesity
Keywords: insulin therapy; hepatic fat; type 2 diabetes; body composition; comparison of insulin detemir and insulin glargine; Changes in Hepatic Fat; Obesity
MeSH Terms: conditions — Diabetes Mellitus; Obesity; Diabetes Mellitus, Type 2 | interventions — Insulin Glargine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- insulin Levemir (Experimental)
  Interventions: Drug: insulin Levemir
- insulin Lantus (Experimental)
  Interventions: Drug: insulin Lantus

INTERVENTIONS:
Drug: insulin Levemir — The participant will receive an insulin dose of insulin Levemir at dinner subcutaneously according to a dosing algorithm.
  Arms: insulin Levemir
Drug: insulin Lantus — The participant will receive an insulin dose of the insulin Lantus at dinner subcutaneously according to a dosing algorithm.
  Arms: insulin Lantus

SUMMARY:
The main objective of this clinical trial is to investigate hepatic fat as the primary endpoint along with body fat, and weight changes after initiation of a basal insulin therapy together with data acquisition that is today's standard in studies investigating obesity and eating patterns with insulin detemir and insulin glargine.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years and < 80 years
* Gender: female, male
* Type 2 diabetes
* BMI: 20.0 - 38.0
* Anti-GAD antibody negative
* Fasting blood glucose > 126 mg/dl
* HbA1c 7.0 - 11.0%
* Need for insulin therapy

Exclusion Criteria:

* Previous therapy with insulin within the last 3 months prior to inclusion into the study
* Previous therapy with glitazones within the last 6 months prior to inclusion into the study
* Change in therapy with lipid-lowering or anti-hypertensive agent within one month prior to inclusion into the study (a stable lipid-lowering or anti-hypertensive therapy is allowed)
* Concomitant participation in other clinical trials
* Type 1 diabetes
* Cardiac and macrovascular disease
* Malignancy including leukaemia and lymphoma within the last 5 years
* Liver disease: cirrhosis or chronic active hepatitis, except fat liver
* Significant renal dysfunction
* other Endocrine disease
* significant laboratory abnormalities
* History of active substance abuse (including an average alcohol consume of > 40g/day and drugs) within the past 2 years
* Female patients: Pregnancy or childbearing potential without adequate contraception (for male patients contraception is not considered as medically important)
* Present therapy with systemic steroids
* Presence of psychiatric disorder or intake of anti-depressive or anti-psychotic agents with the exception of benzodiazepines and SSRIs/SNRI´s
* Use of anti-obesity drugs 3 months prior or during the trial
* Potentially unreliable subjects, probably non compliant subjects, and those judged by the investigator to be unsuitable for the study
* Contraindications for MRI scanning such as persons with cardiac pacemaker and implants out of metal or claustrophobia
* Known hypersensitivity to insulin detemir, insulin glargine or to any of the other components

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2007-11

PRIMARY OUTCOMES:
To describe changes in hepatic fat content between groups. | week 26, week 52

SECONDARY OUTCOMES:
To describe the weight changes from baseline to month 12 between the groups following a subcutaneous treatment strategy with either insulin detemir or insulin glargine. | week 26, week 52
To evaluate changes in body fat and visceral adipose tissue between groups. | week 26, week 52
To describe changes in waist and hip circumferences between groups. | weel 26, week 52
To describe changes in eating behavior and food selection between groups. | week 26, week 52
To describe changes in well being and disease perception between groups. | week 26, week 52
To evaluate the daily insulin dose between groups. | 1 year
To describe the fasting blood glucose between groups. | 1 year
To evaluate hypoglycaemia between groups. | 1 year
To evaluate safety between groups. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Fritsche, Prof. Dr., Principal Investigator — University Hospital of Tübingen; Hermann Toplak, Prof. Dr., Principal Investigator — University Hospital Graz; Peter Diem, Prof. Dr., Study Chair — Bern University Hospital; Alexandra Kautzky-Willer, Prof. Dr., Study Chair — Medical University Vienna; Thomas Pieber, Univ. Prof. Dr., Principal Investigator — Medical University of Graz
Locations (5):
- Austria (3):
  - Medical University Graz, Graz
  - University Hospital Graz, Graz
  - Medical University Vienna, Vienna
- University Hospital of Tübingen, Tübingen, Germany
- University Hospital, Bern, Switzerland